CLINICAL TRIAL: NCT06859086
Title: Clinical Evaluation of Self- Cure Bulk-Fill Resin Composite Versus Conventional Bulk-Fill Resin Composite in Restoration of Proximal Lesions Over a Period Of 24 Months Follow-Up: A Randomized Clinical Trial
Brief Title: Clinical Evaluation of Self- Cure Bulk-Fill Resin Composite Versus Conventional Bulk-Fill Resin Composite Versus Conventional Bulk-Fill Resin Composite Clinical Evaluation of Self- Cure Bulk-Fill Resin Composite Versus Conventional Bulk-Fill Resin Composite
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Wafaa Marei Kakat, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SELF- CURE BULK-FILL RESIN
Record Dates: First submitted 2025-02-23; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Proximal Cavities of Posterior Teeth

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self- Cure Bulk fill Resin Composite (Stela Automix or Stela Capsule, SDI Ltd, Australia) (Experimental): New (Stela, SDI Ltd, Australia) restorative Self-cure: using the stela primer then stela composite with no curing.
  Interventions: Procedure: class II restoration
- Bulk-fill Resin Composite. (Tetric N-Ceram Bulk Fill, Liechtenstein) (Active Comparator): After selective etching of enamel and bonding, the bulk-fill composite resins are inserted then curing.
  Interventions: Procedure: class II restoration

INTERVENTIONS:
Procedure: class II restoration — A class II cavity will be prepared after local anesthesia has been given as requierd . Rubber dam isolation will be done. Sectional matricing and wedging will be done. Followed by placement of restorative material according to the randomization sequence.

SUMMARY:
the aim of this study is To evaluate and compare the clinical performance of Self- Cure Bulk fill Composite Resin Versus Conventional Bulk fill resin composite in Restoration of Proximal Lesions over a Period of 24 months Follow-up.

DETAILED DESCRIPTION:
Examination and selection of all patients will be done according to inclusion and exclusion criteria. A class II cavity will be prepared after local anesthesia has been given as required. Sectional matricing and wedging will be done.Followed by, placement of restorative material according to the randomization sequence.

For the intervention: The sectional matrix will be applied first, followed by filling of cavity with Self-Cure bulk-fill Resin Composite. (Stela Automix or Stela Capsule, SDI Ltd, Australia) For the control group: The sectional matrix will be applied first, followed by filling of the cavity with the bulk-fill resin composite material (Tetric N-Ceram Bulk Fill, Liechtenstein). Clinical evaluation will be done using USPHS criteria at 6,12,18 and 24 monthes follow up

ELIGIBILITY:
Patient-related criteria:

Inclusion criteria:

* Patients consulting in one of the outpatient clinics listed above.
* Able to tolerate necessary restorative procedures.
* Provide informed consent.
* Accepts the 18 months follow-up period.

Exclusion criteria:

* Medically compromised patients, as they will not be able to attend multiple appointments or may require special management.
* Pregnant women; as radiographs cannot be taken for them.
* Allergy to any of the restorative materials, including anesthetics.
* Uncooperative patients, will not abide by the instructions or attend the appointments.

Tooth related criteria:

Inclusion criteria:

* Teeth with primary proximal carious lesions.
* Teeth are vital according to pulp-sensitivity tests.
* Well-formed and fully-erupted in normal functional occlusion with natural antagonist and adjacent teeth.

Exclusion criteria:

* Deciduous teeth; as the study is targeting only permanent teeth.
* Teeth with previous restorations, which may add another variable to the study (type of old restorative material, extent of recurrent caries).
* Spontaneous pain or prolonged pain after sensitivity tests (cold and electrical tests), which would indicate irreversible pulpal damage.
* Negative sensitivity tests, periapical radiolucencies and sensitivity to axial or lateral percussion, which would indicate pulp necrosis.
* Teeth presenting external or internal resorption, with adverse pulpal reactions which may affect the outcome of the study.
* Teeth with cervical caries; which can't be evaluated on periapical radiographs.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Marginal adaptation | 24 months
  The restoration will be clinically assessed using USPHS criteria. Restoration will be given Alpha for the ideal clinical situation, Bravo for acceptable and charlie for clinically unacceptable and in need of replacement.

SECONDARY OUTCOMES:
Marginal discoloration | 24 months
  The restoration will be clinically assessed using USPHS criteria. Restoration will be given Alpha for the ideal clinical situation, Bravo for acceptable and charlie for clinically unacceptable and in need of replacement.
Recurrent caries | 24 months
  The restoration will be clinically assessed using USPHS criteria. Restoration will be given Alpha for the ideal clinical situation and charlie for clinically unacceptable and in need of replacement.
Retention analysis | 24 months
  The restoration will be clinically assessed using USPHS criteria. Restoration will be given Alpha for the ideal clinical situation and charlie for clinically unacceptable and in need of replacement.
Surface roughness | 24 months
  The restoration will be clinically assessed using USPHS criteria. Restoration will be given Alpha for the ideal clinical situation, Bravo for acceptable and charlie for clinically unacceptable and in need of replacement.
Postoperative sensitivity | 24 months
  The restoration will be clinically assessed using USPHS criteria. Restoration will be given Alpha for the ideal clinical situation and charlie for clinically unacceptable and in need of replacement.
Anatomic form | 24 months
  The restoration will be clinically assessed using USPHS criteria. Restoration will be given Alpha for the ideal clinical situation, Bravo for acceptable and charlie for clinically unacceptable and in need of replacement.
Proximal contact | 24 months
  The restoration will be clinically assessed using USPHS criteria. Restoration will be given Alpha for the ideal clinical situation, Bravo for acceptable and charlie for clinically unacceptable and in need of replacement.
Color match | 24 months
  The restoration will be clinically assessed using USPHS criteria. Restoration will be given Alpha for the ideal clinical situation, Bravo for acceptable and charlie for clinically unacceptable and in need of replacement.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided